CLINICAL TRIAL: NCT03539432
Title: Exploration of Gemfibrozil as a Treatment for Alcohol Use Disorder
Brief Title: Exploration of Gemfibrozil as a Treatment for AUD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funds for the study expired
Sponsor: The Mind Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-018
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Results first posted 2021-10-18 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-09

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Gemfibrozil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gemfibrozil (Experimental): Gemfibrozil 600 mg by mouth twice daily
  Interventions: Drug: Gemfibrozil 600 MG
- Placebo (Placebo Comparator): Microcrystalline cellulose powder packaged in capsules identical to the experimental condition
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Gemfibrozil 600 MG — Gemfibrozil capsules (600 mg) taken twice per day
  Arms: Gemfibrozil
Drug: Placebo oral capsule — Microcrystalline cellulose powder packaged in capsules identical to the experimental medication
  Arms: Placebo

SUMMARY:
This study will examine the efficacy of the medication gemfibrozil in reducing alcohol consumption in individuals with an alcohol use disorder who are seeking treatment for alcohol-related problems. Twenty individuals will be randomized to receive four weeks of either gemfibrozil or placebo and retrospective reports of alcohol use will be collected throughout the trial. In addition, brain imaging measures will be collected at baseline and after two weeks of treatment to determine the effects of gemfibrozil on brain functioning.

ELIGIBILITY:
Inclusion Criteria:

1. males and females age 18-60 meeting DSM-V criteria for moderate or severe AUD in the past year
2. interested in cutting down or quitting drinking
3. able to provide voluntary informed consent
4. have at least 4 heavy drinking days (≥ 5 drinks per day for men, and 4 for women) in the past 30 days

Exclusion Criteria:

1. severe liver disease; severe kidney disease; gallbladder disease or gallstones
2. chronic renal or hepatic failure
3. recent pancreatitis
4. insulin-dependent diabetes
5. other urgent medical problems
6. moderately elevated liver function tests (AST or ALT greater than 2 times upper limit of normal) or elevated creatine kinase (CK)
7. schizophrenia, schizoaffective disorder, Bipolar I disorder, suicidal thoughts in the last month
8. current moderate or severe other substance use disorder (SUD; except nicotine or marijuana)
9. active legal problems with the potential to result in incarceration
10. pregnancy or lactation, or child bearing age and not on birth control or not willing to use other birth control methods (e.g. condoms)
11. current daily use of anti-craving medications, mood stabilizers, benzodiazepines, or anti-psychotics
12. regularly taking a medication contraindicated for use with gemfibrozil including other fibrates, statins, repaglinide, or which are believed to interact with gemfibrozil such as dasabuvir, dabrafenib, loperamide, montelukast, paclitaxel, pioglitazone, rosiglitazone, colestipol, colchicine and warfarin41,68
13. a history of alcohol withdrawal-induced seizures or delirium tremens (hallucinations, disorientation) requiring hospital admission during the last ten years
14. a history of moderate or severe traumatic brain injury (TBI; loss of consciousness >30 minutes69)
15. left-handedness
16. any contraindications for MRI

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Mind Research Network, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemfibrozil | Placebo
Started | 2 | 1
Completed | 2 | 0
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemfibrozil | Placebo | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Standard Drinks Per Drinking Day
Description: Average number of standard drinks consumed on drinking days
Time Frame: Baseline
Measure: Mean (Full Range); unit: Drinks per drinking day
Arm/Group | Gemfibrozil | Placebo
Number analyzed (Participants) | 2 | 1
Drinks per drinking day | 6.17 [5.57 to 6.76] | 8.59 [8.59 to 8.59]

2. Primary Outcome: Mean Standard Drinks Per Drinking Day
Description: Average number of standard drinks consumed on drinking days
Time Frame: 2 weeks post baseline
Population: The one participant in the placebo condition dropped out before taking any medication
Measure: Mean (Full Range); unit: Drinks per drinking day
Arm/Group | Gemfibrozil | Placebo
Number analyzed (Participants) | 2 | 0
Drinks per drinking day | 4.12 [3.58 to 4.667] |

3. Primary Outcome: Mean Standard Drinks Per Drinking Day
Description: Average number of standard drinks consumed on drinking days
Time Frame: 4 weeks post baseline
Population: The one participant in the placebo condition dropped out before taking any medication
Measure: Mean (Full Range); unit: Drinks per drinking day
Arm/Group | Gemfibrozil | Placebo
Number analyzed (Participants) | 2 | 0
Drinks per drinking day | 2.18 [2 to 2.35] |

4. Primary Outcome: Percent Days Abstinent
Description: Percentage of days of abstinence from alcohol
Time Frame: Baseline
Measure: Mean (Full Range); unit: Percentage of abstinent days
Arm/Group | Gemfibrozil | Placebo
Number analyzed (Participants) | 2 | 1
Percentage of abstinent days | 31 [16.7 to 44.4] | 32.2 [32.2 to 32.2]

5. Primary Outcome: Percent Days Abstinent
Description: Percentage of days of abstinence from alcohol
Time Frame: 2 weeks post baseline
Population: The one participant in the placebo condition dropped out before taking any medication
Measure: Mean (Full Range); unit: Percentage of abstinent days
Arm/Group | Gemfibrozil | Placebo
Number analyzed (Participants) | 2 | 0
Percentage of abstinent days | 45.5 [0 to 90.9] |

6. Primary Outcome: Percent Days Abstinent
Description: Percentage of days of abstinence from alcohol
Time Frame: 4 weeks post baseline
Population: The one participant in the placebo condition dropped out before taking any medication
Measure: Mean (Full Range); unit: Percentage of abstinent days
Arm/Group | Gemfibrozil | Placebo
Number analyzed (Participants) | 2 | 0
Percentage of abstinent days | 45 [0 to 90] |

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Gemfibrozil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/2 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemfibrozil (N=2) | Placebo (N=1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (Nervous system disorders) | 1 (1) | 0 (0)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT03539432/Prot_SAP_002.pdf
  • Informed Consent Form (2018-06-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT03539432/ICF_003.pdf